CLINICAL TRIAL: NCT03920371
Title: Extended Pilot Evaluation of a Prototype Hand Held Hybrid Gamma Camera
Brief Title: Evaluation of a Prototype Hand Held Hybrid Gamma Camera
Acronym: BIVISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0591
Record Dates: First submitted 2017-01-16; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-05

CONDITIONS: Tumour
Keywords: small field of view; hybrid compact gamma camera; handheld gamma camera
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gamma camera imaging (Experimental): hand held camera
  Interventions: Other: gamma camera imaging

INTERVENTIONS:
Other: gamma camera imaging — Following the administration of the routine radiopharmaceutical and the standard wait before clinical diagnostic imaging, additional research gamma camera imaging is carried out

SUMMARY:
The aim of the project is to undertake clinical development of a hybrid compact gamma camera that combines gamma ray and optical imaging. It is an extension of the previous pilot study using a newly developed handheld hybrid compact gamma camera in clinical arena.

DETAILED DESCRIPTION:
This is a single visit study involving patients who have been referred to the Nuclear Medicine Clinic at Nottingham University Hospitals as part of a standard diagnostic test. Each patient's participation will be approximately 30 minutes and not normally longer than one hour. The study will run for 11 months commencing February 2017 and ceasing at the end of December 2017.

As part of their routine care, patients will be sent a letter booking their diagnostic test through a Nuclear Medicine Clinic. Once they have confirmed that they will be attending this diagnostic test, one of the clinical study team trained to take consent will contact the patient by phone. At this point they will be informed of the reason for the study, why they have been approached and the study schedule. If they express interest in participating they will then be sent a copy of the patient informed consent forms. They will be given a minimum of 24 hours before formally signing consent at the study site immediately before participating.

Study plan:

Following the administration of the routine radiopharmaceutical and the standard wait before clinical diagnostic imaging, the patient will have research images acquired using the hybrid prototype gamma camera. All research images will be anonymised and the additional imaging performed as part of this study will fit in with the patient and the diagnostic test schedules. Should the patient wish to stop at any point, the research study procedure will be terminated. Once these images have been acquired then the patient will go home or proceed with the requirements of their diagnostic test. 75 participants will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study;
* Male or Female, aged 18 years or above;
* Be able to understand the study, willing to co-operate with the study procedures and able to attend the study assessment;
* Have been administered a radiopharmaceutical as part of a diagnostic test.

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the study;
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study;
* Patients who have had a nuclear medicine procedure with administration of a radiopharmaceutical within 72 hours prior to the procedure.
* Patients who do not speak or understand English (since no translator will be available).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Agreement of the visualisation of radiopharmaceutical uptake between the hybrid gamma camera and the standard clinical gamma camera for the sites investigated. | 1 year
  The subjective assessment of scintigraphic images obtained using the hybrid camera under test and the standard clinical gamma camera.
  The image data will be didvdiid into the different exam types and scored using a 3 point scale.

SECONDARY OUTCOMES:
The clinical optimisation of the hybrid gamma camera image display | 1 year
  Following subjective assessment of the recorded images the data set will be reviewed by experienced observers and the display fusion will be modified to obtain the clearest visualisation of radiopharmaceutical uptake.

CONTACTS AND LOCATIONS:
Overall Officials: John E Lees, PhD, Study Director — University of Leicester
Locations (1):
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng AH, Clay D, Blackshaw PE, Bugby SL, Morgan PS, Lees JE, Perkins AC. Assessment of the performance of small field of view gamma cameras for sentinel node imaging. Nucl Med Commun. 2015 Nov;36(11):1134-42. doi: 10.1097/MNM.0000000000000377. PMID 26352214
- [Background] Bugby SL, Lees JE, Bhatia BS, Perkins AC. Characterisation of a high resolution small field of view portable gamma camera. Phys Med. 2014 May;30(3):331-9. doi: 10.1016/j.ejmp.2013.10.004. Epub 2013 Nov 10. PMID 24225012
- [Background] Bhatia BS, Bugby SL, Lees JE, Perkins AC. A scheme for assessing the performance characteristics of small field-of-view gamma cameras. Phys Med. 2015 Feb;31(1):98-103. doi: 10.1016/j.ejmp.2014.08.004. Epub 2014 Nov 13. PMID 25440940
- [Background] Lees, J.E., S.L. Bugby, B.S. Bhatia, L.K. Jambi, M.S. Alqahtani, W.R. McKnight, A.H. Ng, and A.C. Perkins, A small field of view camera for hybrid gamma and optical imaging. Journal of Instrumentation, 2014. 9(12): p. C12020-C12020.